CLINICAL TRIAL: NCT06145594
Title: Ecological Momentary Assessment-Guided Transcranial Magnetic Stimulation Maintenance Therapy for Prevention of Depression Relapse or Recurrence
Brief Title: EMA-Guided Maintenance TMS for Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1503374
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial Magnetic Stimulation (TMS); Ecological Momentary Assessment (EMA); Major Depressive Disorder (MDD); Maintenance Therapy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Randomized, 2 parallel groups (EMA or EMA+mTMS) with longitudinal follow-up (with EMA monitoring) over 1 year. open-label mTMS and other concurrent treatment as usual (TAU) for bother groups; Adjunct mTMS is offered if/when determined by software algorithm for EMA+mTMS group only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMA+Maintenance TMS (Experimental): Weekly EMA monitoring and a cluster of 5 maintenance sessions scheduled if/when PHQ9 scores reach threshold, per algorithm. Participants continue other concurrent treatment as usual (TAU) with medications, psychotherapy, etc per outpatient clinicians.
  Interventions: Other: EMA Monitoring; Other: Scheduling Maintenance TMS sessions
- EMA only (Active Comparator): Weekly EMA monitoring without scheduled maintenance TMS. Participants in this arm may get TMS retreatment according to current standard of care (i.e., through their insurance coverage). Participants continue other concurrent treatment as usual (TAU) with medications, psychotherapy, etc per outpatient clinicians.
  Interventions: Other: EMA Monitoring

INTERVENTIONS:
Other: EMA Monitoring — Weekly prompts to participants' smart phones for collection of PHQ-9 data
Other: Scheduling Maintenance TMS sessions — When threshold score is reached, the participants is offered TMS maintenance treatments
  Arms: EMA+Maintenance TMS

SUMMARY:
The goal of this study is to evaluate the use of ecological-momentary-assessment (EMA) as a method for scheduling maintenance treatments for patients with Major Depressive Disorder (MDD) who responded to an initial acute course of Transcranial Magnetic Stimulation (TMS). To assess symptom re-emergence and severity over time, the Patient Health Questionnaire-9 item (PHQ-9) will be administered weekly via a prompt with a link send to a participants' smart phones. Adaptive algorithm software will monitor each participant's PHQ-9 scores over time and determine when a threshold increase in symptoms has occured and maintenance TMS sessions should be offered. Participants in this study will be randomized to either receive weekly EMA (monitoring only) or weekly EMA with maintenance TMS sessions (scheduled as indicated by the EMA algorithm). Participation for each subject will last for one year, with maintenance TMS offered as an adjunct to ongoing treatment as usual (TAU) for depression, i.e., ongoing pharmacotherapy, psychotherapy.

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS or simply '"TMS") is a FDA approved non-invasive treatment modality for treatment-resistant MDD. While the current standard of care defines the treatment schedule for an acute course (i.e., 30 sessions delivered once daily over 6 weeks, followed by several weeks of sessions in a taper schedule), there is no current standard for scheduling maintenance TMS sessions to keep patients well after they have completed an initial course of TMS Therapy. Several prospective studies show that re-introduction of TMS is highly successful for rescuing patients who have MDD symptom relapse, but those trials used serial assessment of depressive symptoms at regular intervals over time and applied specific criteria for triggering the re-introduction of TMS treatments - a method which has not been translated to real-life clinical practice.

Follow-up data show TMS responders are highly variable with regard to how long they will sustain their benefits after completing the course of TMS; some will sustain response/remission for years while others will relapse after weeks or months. One randomized prospective study that aimed to prevent depressive episode relapse with maintenance TMS showed that a fixed (once per month) treatment schedule was not better than "watchful waiting" with threshold symptom-triggered TMS sessions. It is clear that there is not a "once size fits all" treatment schedule that should be applied for TMS maintenance therapy. Considering the wide range in durability of effect, a personalized approach is needed for determining when TMS maintenance treatments should be given. This study evaluates a convenient method for monitoring symptoms over time and a customized approach to scheduling maintenance TMS sessions on an individual-patient basis, with the "trigger" for re-introduction of TMS treatments driven by patient-specific change in MDD symptoms.

Ecological Momentary Assessment (EMA) involves measurement of symptoms in the real-life daily environment in which a patient lives, works, and functions, rather than in the research or clinic setting. One popular method for EMA involves using applications that are downloaded to a patient' smart phone or cloud-based software platforms which can sed a text message prompt to the patient at pre-set times so the patient can report about their symptoms. This study will evaluate whether a method that uses EMA assessments (weekly PHQ-9 surveys) and adaptive algorithm software can be used to schedule maintenance TMS sessions for MDD patients who have responded to a standard acute course of TMS therapy.

MDD patients who initially responded to a standard course of TMS at Butler Hospital will be invited to participate in this EMA study. Participants will be prompted to complete a brief symptom scale (PHQ-9) weekly via smart phone prompts. The software will compare their scores each week to a target score set for them (customized for each participant based on their response to the TMS acute course) and also compare the degree of change in their scores from week to week. The EMA software algorithm determines if and when a patient's score reaches a threshold that indicates maintenance TMS sessions may be appropriate.

Participants will be randomized to one of two groups: EMA only (EMA) or EMA with TMS maintenance sessions offered when their scores show a threshold level of increase relative to their "target" score (EMS+mTMS). While we routinely recommend patients avoid abrupt or significant changes to their psychotropic medication regimen following a successful acute course of TMS, both groups will continue to receive treatment as usual (TAU) for their depression in the form of pharmacotherapy or psychotherapy as prescribed or administered by their providers in the community. Other treatments will not be controlled, so mTMS sessions will thus be considered adjunctive therapy for those in the EMA+mTMS group who receive them. mTMS will be delivered as a "cluster" of 5 TMS sessions over 3-5 days, and will be offered only when there threshold level of MDD symptom re-emergence. Response to a cluster of maintenance sessions will also be assessed by EMA, with PHQ-9 surveys delivered at fixed intervals (2 days and 4 days) after the final session in the mTMS cluster is delivered.

The mTMS sessions will be delivered as standard-of-care, evidence-based protocols, with the selection of protocol for each session determined by TMS-trained treating physicians and based on consideration the patient's history of prior TMS response and tolerability, patient preference, etc. When two sessions are delivered in the same day, there will be a rest period of 45 minutes between each session.

Both EMA and EMA+mTMS groups will complete assessments by phone every 3 months to collect data about use of medications and utilization of other treatments. Patients in either group who experience significant MDD symptom relapse and meet coverage criteria for TMS re-treatment according to their health insurance policy may be referred for a standard insurance-covered TMS re-treatment course at any time during their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary Major Depressive Disorder who responded (50% drop in score from pre-treatment baseline to final score on depression scale) to a standard acute course of TMS Therapy at Butler Hospital.
* PHQ-9 <10
* Must have access to smart phone and ability to use electronic device
* Continues to meet standard eligibility criteria for clinical TMS procedures and have been medically cleared to receive treatments, per physician judgement.

Exclusion Criteria:

•Per physician judgement: Meets standard clinical exclusion criteria for TMS based on safety, e.g., seizure disorder, significant brain injury/intracranial mass, implanted ferromagnetic metal within 30mm of the TMS coil, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Weeks in Response Range | 1 year
  Number of weeks that participants' PHQ-9 total scores remained in their "response" range (equal to or less than their customized PHQ-9 target score+4)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Carpenter, MD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No